CLINICAL TRIAL: NCT07179887
Title: Remote Ischaemic Conditioning in the Older Person and Effects on Dynamic Cerebral Autoregulation
Acronym: RICE-DCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of Leicester (Other)
Responsible Party: Principal Investigator, Timothy England, Professor of Stroke Medicine, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: FMHS 192-0625
Record Dates: First submitted 2025-09-03; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Autoregulation; Blood Pressure; Dynamic Cerebral Autoregulation
Keywords: Remote Ischaemic Conditioning; Dynamic Cerebral Autoregulation; Vascular Health; Randomised Controlled Trial

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose RIC (Experimental): Daily sessions of RIC for 6 weeks. Each session will consist of 4 x 5 minute cuff inflation to 20mmHg above systolic blood pressure, interspersed with 5 minute periods of cuff deflation
  Interventions: Device: Remote Ischaemic Conditioning
- Low dose RIC (Experimental): 3x weekly sessions of RIC for 6 weeks. Each session will consist of 4 x 5 minute cuff inflation to 20mmHg above systolic blood pressure, interspersed with 5 minute periods of cuff deflation
  Interventions: Device: Remote Ischaemic Conditioning
- Sham RIC (Placebo Comparator): 3x weekly sessions of Sham RIC for 6 weeks. Each session will consist of 4 x 5 minute cuff inflation to 20mmHg only, interspersed with 5 minute periods of cuff deflation
  Interventions: Device: Sham Remote Ischaemic Conditioning

INTERVENTIONS:
Device: Remote Ischaemic Conditioning — Cuff inflation to 20mmHg abocve systolic blood pressure for cycles of 5 minutes. Each session will consist of 4 cycles of 5 minte inflation followed by 5 minute deflation. Total session time 40 minutes
  Arms: High dose RIC; Low dose RIC
Device: Sham Remote Ischaemic Conditioning — Cuff inlfation to 20mmHg only for cycles of 5 minutes. Each session will consist of 4 cycles of 5 minute inflation followed by 5 minutes of deflation. Total session time of 40 minutes
  Arms: Sham RIC

SUMMARY:
Remote Ischaemic Conditioning (RIC) is the process of inducing short periods of ischaemia in a limb with the aim of improving vascular health systemically. Recent findings have demonsatrated efficacy in a variety of clinical settings. However, the ideal protocol of RIC [dose] is unknown. Dynamic Cerebral Autoregulation (dCA) has been shown to increase in response to RIC.

The goal of this trial is to study whether an increase in RIC protocol intensity results in a larger effect on biomarkers of vascular health such as dCA.

Participants shall:

Receive RIC daily, RIC thrice weekly or sham RIC thrice weekly for 6 weeks Visit the School of Medicine at baseline and at 6 weeks for measurement of biomarkers of vascular health including blood pressure, indices od dCA and blood plasma samples

DETAILED DESCRIPTION:
Remote Ischaemic Conditioning (RIC) involves the delivery of short periods of ischaemia to a limb (using a blood pressure cuff), with the aim of promoting resilience to ischaemia in distant organs. It has shown promise as in intervention in both the treatment of acute ischaemic stroke and secondary prevention of cerebrovascular events. Various protocols exist ranging from single sessions of RIC delivered around the time of an ischaemic event, known as acute RIC, to repeated sessions delivered over days, weeks or even months, known as chronic RIC.

Preclinical work in animal models of stroke demonstrated consistent benefits of RIC. However, translation of these findings to human trials has yielded mixed results. Two large randomised controlled trials conducted in recent years have suggested benefit where RIC is given as a treatment following acute ischaemic stroke or when used in the secondary prevention of stroke in patients with symptomatic intracranial atherosclerosis. However, other clinical trials of RIC have yielded neutral results. For example, the RESIST trial, which used RIC as an intervention following both acute ischaemic and haemorrhagic stroke.

It is not known exactly why the promising findings in preclinical studies have not been replicated in human trials. It is likely that protocols of RIC, i.e. the 'dose', which proved effective in animal models of stroke, may not be sufficient when applied to multimorbid human populations who have also received current standard therapy. These therapies, such as antiplatelets, themselves provide cerebrovascular protection and may abrogate some of the benefit of RIC. It may be that more intense protocols of RIC, particularly chronic RIC, are needed to illicit benefit in humans.

To answer this question, work should be done to investigate the effect of RIC protocol intensity on vascular health in older adults. Too often in RIC research, there has been a rapid jump from preclinical study to large RCT. These RCTs initially used protocols of RIC based on those used in preclinical studies. With increasing awareness of the potential problems with this approach, RCTs now tend to use more intense protocols of RIC. However, very little work has been done examining the effect of RIC on biomarkers of vascular health to inform the choice of RIC dose, informing future trial design.

Dynamic cerebral autoregulation (dCA) is a measure of the regulation of cerebral blood flow in response to changes in systemic blood pressure. It has been shown to be impaired in the immediate post stroke period (≈2 weeks) and severely impaired autoregulation in the hours after stroke has been correlated with worse outcomes. Dynamic Cerebral Autoregulation has also been shown to improve in young adults given 2 weeks of RIC. We propose to conduct a further study in older adults, aged 65-85, investigating the effect of chronic RIC on biomarkers of vascular health including dCA and blood pressure (BP), comparing two difference dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Participant aged 65 - 85
* Participant is able to perform RIC independently at home

Exclusion Criteria:

* Active cardiovascular or cerebrovascular disease (acute event within the last 12 months)
* Atrial fibrillation or other significant arrhythmias
* Peripheral Vascular Disease
* Haemostatic disorders
* Soft tissue injury or fracture to the upper limb
* Pregnant or breast feeding
* History or current psychiatric illness
* History or current neurological condition (e.g. epilepsy)
* Inability to identify temporal window for transcranial doppler ultrasound at screening visit
* Any condition or presentation under current investigation that is deemed by the study clinician to exclude the participant from the study.
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Autoregulatory Index | Baseline and 6 weeks
  In dynamic cerebral autoregulation analysis, the Autoregulatory Index is a dimensionless index ranging from 0 to 9. 0 represents no autoregulation and 9 represents very strong autoregulation

SECONDARY OUTCOMES:
Phase DIfference | Baseline and 6 weeks
  In dynamic cerebral autoregulation analysis, the phase difference quantifies the timing shift between oscillations in arterial blood pressure (ABP) and cerebral blood flow velocity (CBFV) at a given frequency. It is reported in degrees with higher values representing stronger autoregulation
Gain | Baseline and 6 weeks
  In dynamic cerebral autoregulation analysis, the Gain quantifies the magnitude of transmission of blood pressure oscillations into cerebral blood flow oscillations. It is reported both as cm/s/mmHg. Lower values represent better autoregulation.
Clinic Systolic Blood Pressure | Baseline and week 6
  Resting blood pressure will be calculated using automated sphygmomanometer. The average of 3 recordings will be used. Blood pressure will be rexpressed in units of mmHg.
Clinic Diastolic Blood Pressure | Baseline to 6 Weeks
  Resting blood pressure will be calculated using automated sphygmomanometer. The average of 3 recordings will be used. Blood pressure will be rexpressed in units of mmHg.
Clinic Mean Arterial Pressure | Baseline to 6 Weeks
  Resting blood pressure will be calculated using automated sphygmomanometer. The average of 3 recordings will be used. Blood pressure will be rexpressed in units of mmHg.
Blood plasma markers | Baseline and 6 weeks
  Markers of RIC efficacy will be measured by ELISA from blood plasma stored at the time of data collection and analysed at study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Tim England, MBChB PhD, Principal Investigator — University of Nottingham
Locations (1):
- School of Medicine, University of Nottingham, Royal Derby Hospital Centre, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Bruijn WC, Boeve ER, van Run PR, van Miert PP, Romijn JC, Verkoelen CF, Cao LC, Schroder FH. Etiology of experimental calcium oxalate monohydrate nephrolithiasis in rats. Scanning Microsc. 1994;8(3):541-9; discussion 549-50. PMID 7747156
- [Background] Craft AW. Challenges in the management of bone tumors--1996. Ann N Y Acad Sci. 1997 Sep 17;824:167-79. doi: 10.1111/j.1749-6632.1997.tb46219.x. No abstract available. PMID 9382441
- [Background] Hou C, Lan J, Lin Y, Song H, Wang Y, Zhao W, Li S, Meng R, Hao J, Ding Y, Chimowitz MI, Fisher M, Hess DC, Liebeskind DS, Hausenloy DJ, Huang J, Li Z, Han X, Yang J, Zhou J, Chen P, Zhu X, Hu P, Pang H, Chen W, Chen H, Li G, Tao D, Yue W, Gao Z, Ji X; RICA investigators. Chronic remote ischaemic conditioning in patients with symptomatic intracranial atherosclerotic stenosis (the RICA trial): a multicentre, randomised, double-blind sham-controlled trial in China. Lancet Neurol. 2022 Dec;21(12):1089-1098. doi: 10.1016/S1474-4422(22)00335-0. Epub 2022 Oct 27. PMID 36354026
- [Background] Benedict MQ, McNitt LM, Cornel AJ, Collins FH. A new marker, black, a useful recombination suppressor, In(2)2, and a balanced lethal for chromosome 2 of the mosquito Anopheles gambiae. Am J Trop Med Hyg. 1999 Oct;61(4):618-24. doi: 10.4269/ajtmh.1999.61.618. PMID 10548297
- [Background] Bell RM, Basalay M, Botker HE, Beikoghli Kalkhoran S, Carr RD, Cunningham J, Davidson SM, England TJ, Giesz S, Ghosh AK, Golforoush P, Gourine AV, Hausenloy DJ, Heusch G, Ibanez B, Kleinbongard P, Lecour S, Lukhna K, Ntsekhe M, Ovize M, Salama AD, Vilahur G, Walker JM, Yellon DM. Remote ischaemic conditioning: defining critical criteria for success-report from the 11th Hatter Cardiovascular Workshop. Basic Res Cardiol. 2022 Aug 15;117(1):39. doi: 10.1007/s00395-022-00947-2. PMID 35970954
- [Background] Hougaard KD, Hjort N, Zeidler D, Sorensen L, Norgaard A, Hansen TM, von Weitzel-Mudersbach P, Simonsen CZ, Damgaard D, Gottrup H, Svendsen K, Rasmussen PV, Ribe LR, Mikkelsen IK, Nagenthiraja K, Cho TH, Redington AN, Botker HE, Ostergaard L, Mouridsen K, Andersen G. Remote ischemic perconditioning as an adjunct therapy to thrombolysis in patients with acute ischemic stroke: a randomized trial. Stroke. 2014 Jan;45(1):159-67. doi: 10.1161/STROKEAHA.113.001346. Epub 2013 Nov 7. PMID 24203849
- [Background] Beighton D, Ludford R, Clark DT, Brailsford SR, Pankhurst CL, Tinsley GF, Fiske J, Lewis D, Daly B, Khalifa N, et al. Use of CHROMagar Candida medium for isolation of yeasts from dental samples. J Clin Microbiol. 1995 Nov;33(11):3025-7. doi: 10.1128/jcm.33.11.3025-3027.1995. PMID 8576366
- [Background] Beilman GJ, Cerra FB. The future. Monitoring cellular energetics. Crit Care Clin. 1996 Oct;12(4):1031-42. doi: 10.1016/s0749-0704(05)70291-8. PMID 8902383